CLINICAL TRIAL: NCT06035042
Title: 4P: Persistent Postoperative Pediatric Pain
Acronym: 4P
Status: Completed | Type: Observational
Sponsor: Region Halland (Other)
Collaborators: Lund University (Other); Region Skane (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Anna Persson, Consultant in Anaesthesia and Intensive Care Medicine, PhD, Region Halland
Other Study IDs: 2022-04821
Record Dates: First submitted 2023-05-29; First posted 2023-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: Pediatric pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Scheduled surgery — All subjects will be exposed to surgery

SUMMARY:
For children, adequate perioperative pain management is a right according to the UN convention on the rights of the child, a law in Sweden since 2020. Despite this, children are still under-treated in many cases. In addition to great suffering, this can lead to missing school and a long-term burden on the society.

ESPA, the European Society for Pediatric Anesthesia, has drawn up guidelines for perioperative pain management. With the study 4P: Persistent Postoperative Pediatric Pain, we want to investigate whether these guidelines are followed and how many children develop long-term pain postoperatively.

In order to map the prevalence of pain after surgery in children in Sweden, the investigators plan to include and follow 2000 children in southern Sweden who undergo surgery. The study provides a unique opportunity to follow a large number of children, evaluate given per- and postoperative pain treatment and identify factors linked to the development of acute and long-term postoperative pain. Our goal is to optimize peri- and postoperative pediatric pain management to promote rapid recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-17 years
* Scheduled surgery for hernia, penile surgery, retentio testis, adenotonsillectomy, appendectomy or acute fracture in southern Sweden.
* Informed consent

Exclusion Criteria:

* Scheduled for several surgeries within the time-frame
* Inability to understand swedish
* Inability to understand the meaning of participation.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with planned surgery in southern Sweden for by ESPA specified types of surgeries.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Incidence of acute postoperative pain | Within 24 hours after surgery
  How many children experience acute postoperative pain after surgery in Sweden?
Adherence to guidelines from ESPA regarding perioperative analgesia | Perioperative
  How many patients are treated according to the suggested guidelines regarding pain treatment from ESPA (%)? Do they experience less postoperative pain (FLACC/FPS/NRS 0-10)? Groups compared with MannWhitney U-test. Also description of the deviation.
Incidence of persistent postoperative pain | At 3 months after surgery
  How many children experience persistent postoperative pain after surgery in Sweden?
Incidence of persistent postoperative pain | At 6 months after surgery
  How many children experience persistent postoperative pain after surgery in Sweden?
Incidence of persistent postoperative pain | At 1 year after surgery
  How many children experience persistent postoperative pain after surgery in Sweden?

SECONDARY OUTCOMES:
Do regional blocks influence the level of acute postoperative pain? | Acute - within 24 hours.
  Do children who recieve a regional block experience less postoperative pain? Croups compared with MannWhitney U-test.
Do regional blocks influence the level of persistent pain? | 3 months after surgery
  Do children who recieve a regional block experience less postoperative pain? Croups compared with MannWhitney U-test.
Parental stress | Within 24 hours
  Does the subjective level of stress, measured on a scale from 0-10 by the parents, affect the experience of acute postoperative pain? Correlation between pain (FLACC/FPS/NRS depending on age) correlated to subjective stress using Spearman Rho.
Parental stress | 3 months after surgery
  Does the subjective level of stress, measured on a scale from 0-10 by the parents, affect the experience of persistent postoperative pain? Correlation between pain (FLACC/FPS/NRS depending on age) correlated to subjective stress using Spearman Rho.
Age | Acute (24 hours) and persistent (3,6 months and 1 year)
  Which age-groups experience most pain. Pain evaluated with FLACC/FPS/NRS depending on age. Risk evaluated with logistic regression.
Gender | Acute (24 hours) and persistent (3,6 months and 1 year)
  Do girls experience more pain than boys? Pain evaluated with FLACC/FPS/NRS depending on age. Risk evaluated with logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Anna KM Persson, MD, PhD, Principal Investigator — Region Halland
Locations (4):
- Sweden (4):
  - Queen Silvias Childrens Hospital Sahlgrenska University Hospital, Gothenburg
  - Hallands Hospital Halmstad, Halmstad
  - Helsingborgs Hospital, Helsingborg
  - Lund childrens hospital, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broman J, Nielsen N, Persson AKM. A prospective observational study on persistent postoperative pediatric pain, 4P: The study protocol. PLoS One. 2025 Jan 14;20(1):e0316533. doi: 10.1371/journal.pone.0316533. eCollection 2025. PMID 39808613